CLINICAL TRIAL: NCT04184037
Title: A Pilot Randomized Controlled Trial of an At-home Mindfulness Meditation Intervention in Older Adults With Mild Cognitive Impairment and in Family Caregivers
Brief Title: iMeditate at Home for Older Adults With Mild Cognitive Impairment and Caregivers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study recruitment was suspended due to interruption of in-person testing after the start of the COVID19 pandemic in March 2020. The current study's protocol is being revised to be delivered fully remotely.
Sponsor: Baycrest (Other)
Collaborators: Center for Aging and Brain Health Innovation (Unknown); InteraXon, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Allison B. Sekuler, Sandra A Rotman Chair in Cognitive Neuroscience; Managing Director and Senior Scientist, Rotman Research Institute; Managing Director, Centre for Aging + Brain Health Innovation; Vice-President Research, Baycrest Health Sciences, Baycrest
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: REB #18-34
Record Dates: First submitted 2019-10-02; First posted 2019-12-03 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Mild Cognitive Impairment; Caregivers
Keywords: Mindfulness meditation; stress reduction; mobile application
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Alprostadil

STUDY DESIGN:
Intervention Model Description: This is a pilot randomised, controlled trial conducted in two study populations: older adults diagnosed with mild cognitive impairment (MCI) and family caregivers of individuals diagnosed with any neurodegenerative disease or MCI. Dyads of participants (older adult with MCI and their caregiver) may also be enrolled. Participants are randomly allocated to a mindfulness meditation with neurofeedback (NFB) or mindfulness meditation without neurofeedback (no-NFB).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The outcomes assessor and all individuals involved in analyzing data will be blind to the participant's study arm. Only the research assistant who will be introducing participants to their meditation app will be aware of their study arm assignment. Participants will be told that they are randomized into one of two types of meditation programs, but will not be told about the difference in the two programs and will not be told if they are in the main intervention group or the control group. That said, given the nature of auditory neurofeedback, participants in the NFB group will be aware that they are receiving neurofeedback. Participants in the no-NFB group will not be experiencing any neurofeedback and, a priori, they should not be aware that neurofeedback is missing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auditory neurofeedback (NFB) (Experimental): Participants in this arm will meditate with the help of a custom version of the Muse app, which guides users in meditation while providing auditory neurofeedback on their state of mindfulness. Participants will wear the EEG headband and headphones when completing the meditation sessions using the app. The neurofeedback consists of changing weather sounds that are heard against a background soundscape (e.g., a beach or rainforest sound). When a user is in a focused state, the weather in the soundscape is good (e.g., it is quiet or a light breeze can be heard). When a user starts mind-wandering, the weather sounds change for the worse: it begins to rain, the wind gets louder, and there may be thunder. When the user returns to a calm state, the weather sounds quiet down again and only the background soundscape is heard. Participants are asked to pay attention to the weather sounds and to use this feedback to train their mind to remain focused on the present moment.
  Interventions: Behavioral: Mindfulness meditation delivered via a mobile app
- No neurofeedback (no-NFB) (Active Comparator): Participants in this arm will meditate using a custom version of the Muse app that is identical in all respects to the mobile app used by the NFB group, expect that the auditory neurofeedback is not active. Participants will wear the EEG headband and headphones when completing the meditation sessions using the app, but the soundscape during the sessions will only contain the background sounds (e.g., the breach or rainforest scene), without any changes to the weather.
  Interventions: Behavioral: Mindfulness meditation delivered via a mobile app

INTERVENTIONS:
Behavioral: Mindfulness meditation delivered via a mobile app — This is a six-week intervention that requires completing daily meditation sessions at home using a mobile app while wearing a four-channel EEG device (Muse,RRID:SCR_014418) and headphones. Participants are asked to increase their session duration from 5 to 15 minutes over the first 10 sessions, and continue with 15 minutes thereafter. Meditation sessions in both intervention arms consist of listening to a calm soundscape while focusing one's attention on the present moment.
  Prior to starting the intervention, participants are familiarized with the mobile device, EEG headband, and the study app during an onboarding session. In this session, participants listen to four different meditation exercise instructions (e.g., focusing attention on their breath, counting breaths, thinking of meditation akin to training a puppy) that offer them techniques to use during meditation.The transcript of these exercises and a basic guide on how to use the study app and headband are provided.
  Other Names: Muse

SUMMARY:
Individuals diagnosed with mild cognitive impairment (MCI) are at a high risk of developing dementia and are an important target population for interventions that may reduce the risk of cognitive decline. A diagnosis of MCI or dementia also has an important impact on caregivers, who show increased levels of stress, anxiety, and depression. Mindfulness meditation is a promising behavioural intervention that may have important benefits both for older adults with MCI and for caregivers. Previous research suggests that meditation may improve psychological wellbeing, reduce stress, and even improve cognitive function. Technology-based mindfulness meditation platforms may be a much-needed solution for promoting the adoption of mindfulness in these populations.

The current study is a pilot randomized control trial of a mindfulness meditation intervention delivered via the Muse platform in two study populations: a) older adults diagnosed with MCI, and b) family caregivers of persons with MCI or neurodegenerative disorders. Muse is a mobile application for meditation that provides real-time feedback about the user's state of mindfulness during meditation via a headband containing electroencephalographic sensors (EEG) that the user wears while meditating. It is thought that this neurofeedback can promote learning and lead to faster improvements in meditation ability and, consequently, greater benefits from meditation practice.

This aim of this pilot study is to establish the acceptability of the Muse platform as an intervention in the two study populations, to determine the feasibility of the randomized control trial designed to evaluate the effectiveness of a 6 week intervention with the Muse platform, and to evaluate the effect of neurofeedback on meditation. Participants will be randomly allocated to meditation with neurofeedback (NFB) or meditation without neurofeedback (no-NFB) and will complete daily meditation sessions for 6 weeks. An assessment visit before and after the intervention will evaluate participants' psychological well-being using questionnaires; their visual working memory, attention, and visual perception using behavioural tests; and their mindfulness ability using questionnaires and a behavioural measure. EEG will also be recorded using the Muse headband to examine changes in electrophysiological markers during cognitive tests and at rest.

DETAILED DESCRIPTION:
The Primary objectives of the main study are:

1. To determine if mindfulness meditation with auditory neurofeedback (NFB) leads to greater improvements in mindfulness relative to a mindfulness meditation without neurofeedback (no-NFB).
2. To determine if a mindfulness meditation intervention with neurofeedback leads to greater improvements in psychological well-being, with perceived stress levels as the primary outcome measure, in the two study populations, relative to a mindfulness meditation program without neurofeedback .

Secondary objectives of the main study are to determine if the NFB intervention leads to greater improvements in 1) other measures of psychological wellbeing and 2 ) behavioural and EEG markers of perceptual and cognitive function, relative to the no-NFB arm, in the two study populations (individuals with MCI; caregivers)

Feasibility and acceptability objectives of the pilot study

1. To evaluate the acceptability of the intervention for older adults with MCI and family caregivers of persons with MCI or neurodegenerative disorders, and to examine whether the acceptability of the intervention is associated with the individual's technological abilities.
2. To estimate the recruitment rate of older adults with MCI and family caregivers separately, as well as dyads of older adults with MCI and their caregivers.
3. To determine the rate of adherence to the intervention schedule (durations per session and number of sessions), and the rate of completion of assessment visits and weekly questionnaires
4. To determine the extent of technical expertise and time resources required of the experimenters to provide technical support to participants in each group
5. To determine the feasibility of blinding experimenters to the intervention arm and of blinding Muse-control participants to the neurofeedback group, given that information about the Muse app is easily available online.
6. To obtain preliminary estimates of the effects of Muse and Muse-control interventions on the psychological well-being, and perceptual and cognitive measures, and the standard deviations of these measures.

Procedures:

Briefly, participants will be enrolled on a continuous basis. After an initial pre-screening phone call or email, interested and eligible participants will come for a consenting and screening visit, which will include a clinical interview to screen for mental-health exclusion criteria, as well as exclusion related to prior use of the Muse device. All those eligible to proceed will return for a baseline assessment visit (Visit 2) where they will complete a series of computer-based task assessments and self-report questionnaires. At the end of the assessments, participants will be introduced to the research assistant responsible for the intervention (training RA). The training RA will train the participant on how to use the Muse headband and app associated with their training condition, as well as give instructions on the required training regimen. The next six weeks will consist of the training period. The training RA will contact participants by phone or email once a week to monitor for any issues. Following the training period, all participants will come back for Visit 3 to repeat the same assessments as were completed at baseline (Visit 2) with the experimenter RAs. All participants will be fully debriefed by the training RA during Visit 3 as to which version of the app they trained with and what the differences are between the two apps.

Sample size justification for the pilot study

A minimum of 12 participants per group and condition is required to provide feasibility and acceptability information. However, to obtain reliable estimates of the variability of each outcome measure, our target sample size is 20 participants per condition (i.e., 40 MCI participants in total and 40 caregivers in total). The actual sample size for the pilot study will be limited by the timeline of the project and the combination of recruitment and retention rates.

Recruitment:

Caregivers will be recruited through advertisements on the Baycrest campus or at institutions that provide services for caregivers. Older adults with MCI will be recruited at Baycrest through advertisements and by contacting eligible participants through the Baycrest Client Registry.

ELIGIBILITY:
Inclusion Criteria (Older adults with MCI):

* Diagnosis of mild cognitive impairment, any type, by a physician at the Baycrest Sam & Ida Ross Memory Clinic
* Confirmation of the absence of progression to dementia within 90 days of study start by a physician or by the study staff
* Aged 55 years to 90 years

Inclusion Criteria (Caregivers):

* Identify as a caregiver of a family member or friend living with mild cognitive impairment (MCI) or any neurodegenerative disease
* Not be financially compensated for their caregiving work
* Aged 20 years to 90 years
* Passes the Telephone Interview for Cognitive Status and Montreal Cognitive Assessment > 23

Exclusion Criteria:

* History of neurological disorders (e.g., malignant brain tumour, multiple sclerosis, Down's syndrome or any other developmental disorders, epilepsy, seizures, Parkinson's, any dementia or neurodegenerative disorder except for MCI), and history of MCI for the caregiver group
* Stroke or history of transient ischemic attack (TIA)
* History of traumatic brain injury (TBI) with loss of consciousness lasting longer than 30 minutes
* Active cancer, history of chemotherapy, or history of radiation to the head
* History of psychiatric conditions including:

  * Diagnosis of major depressive disorder, generalized anxiety disorder, or other psychiatric diagnosis within 90 days of study entry, or
  * Lifetime history of psychosis, bipolar disorder, obsessive compulsive disorder, schizophrenia, or post-traumatic stress disorder
  * History of substance use within the past year
* Serious medical disease that would/could lead to death over the next 2-3 years (e.g. cardiac/renal/liver disease, or cancer) with poor prognosis
* Presence of visual impairment (binocular vision worse than Snellen acuity 20/40)
* Hearing loss that prevents the individual to hear sounds in the Muse app even with a hearing aid (if applicable), or incompatibility of their hearing aid with the Muse headband and inability to hear the Muse app sounds without the hearing aid
* Started taking psychotropic medication (anti-anxiety, anti-psychotics) or cognitive enhancers (memantine, acetylcholinesterase inhibitors) less than 3 months prior to randomization, or has had a change in dosages of any acetylcholinesterase inhibitors or cognitive enhancers within 6 weeks of randomization, or has had any changes in all types of medications or dosages within 4 weeks of randomization.
* Already engages in active meditation practice
* Is enrolled or recently completed (within 30 days) another intervention study or clinical trial
* Unable to understand, read, and speak English

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Change in the Perceived Stress Scale (PSS-10) score | Baseline (Visit 2/Week 1) to Post-Intervention (Visit 3/Week 7).
  The 10-item Perceived Stress Scale is a self-administered questionnaire that measures an individual's perception of how uncontrollable, unpredictable and overloading aspects of their life are on a 5-point scale ranging from 0 (never) to 4 (very often). It has been validated in older adults, caregivers of dementia patients, and dementia patients (Deeken et al., 2018; Ezzati et al., 2014). High scores represent high levels of stress. This is the primary outcome measure in the main study.
Recruitment rate | Study recruitment period, approximately 3 months
  The recruitment rate will be quantified as the number of participants recruited per month, separately for the two study population groups (MCI and caregivers). This is a primary outcome variable for the feasibility study.
Total number of meditation sessions | Intervention period (6 weeks)
  The total number of meditation sessions lasting longer than 3 minutes will be quantified for each participant to evaluate adherence to the intervention schedule. This is a primary acceptability outcome variable for the feasibility study.

SECONDARY OUTCOMES:
Change in breath counting accuracy | Baseline (Visit 2/Week 1), Post-Intervention (Visit 3/Week 7)
  The breath counting task has been proposed and validated as a behavioural measure of mindfulness (Atchley et al., 2016; Levinson et al., 2014; Milz, Faber, Lehmann, Kochi, & Pascual-Marqui, 2014). Participants are asked to breathe normally and count their breaths repeatedly from 1 to 9, pressing one button for counts 1 - 9 and another button for count 9. If the participant loses count, they press a different button to restart the count at 1. A respiration belt will be used to validate the breathing count accuracy.
Change in the Mindfulness Attention and Awareness Scale (MAAS) score | Baseline (Visit 2/Week 1), Post-Intervention (Visit 3/Week 7)
  The MAAS is a 15-item self-administered scale that evaluates the experience of mindfulness in a general, everyday context (Brown & Ryan, 2003). Respondents rate on a six-point scale how frequently they have certain experiences. Higher scores correspond to greater levels of trait mindfulness.
Change in the Perceived Stress Scale (PSS-10) score | Baseline (Visit 2/Week 1) to During Intervention (Week 3)
  The PSS-10 (Cohen et al., 1983) measures an individual's perception of how uncontrollable, unpredictable and overloading aspects of their life are on a 5-point scale ranging from 0 (never) to 4 (very often). The change from baseline to the midpoint of the intervention will be examined to determine the effect over a shorter timespan.
Change in the Beck Depression Inventory (BDI-II) score | Baseline (Visit 2/Week 1), Post-Intervention (Visit 3/Week 7)
  The BDI-II (Steer, Brown, Beck, & Sanderson, 2001) is a 21-item scale scored on a 4-point scale and measures the intensity of self-reported depressive symptoms over the past two weeks, with higher scores representing worse symptoms. The BDI-II has been used with older adults and caregivers of dementia patients (Segal, Coolidge, Cahill, & O'Riley, 2008; Takai et al., 2009)
Change in the Brief Symptom Inventory (BSI) score | Baseline (Visit 2/Week 1), Post-Intervention (Visit 3/Week 7)
  The BSI (Derogatis, 2001) is an 18-item questionnaire that assesses the magnitude of depression, anxiety, and somatic symptoms over the past week using a 5-point scale, from "not at all" to "extremely". The BSI has been used in older adults and caregivers of dementia patients (Anthony-Bergstone et al., 1988; Petkus et al., 2010).
Change in the Warwick Edinburgh Mental Well-being Scale (WEMWBS) score | Baseline (Visit 2/Week 1), Post-Intervention (Visit 3/Week 7)
  The WEMWBS measures mental well-being, with a focus on positive aspects (Tennant et al., 2007). It has 14 items with 5 response categories, summed to a single score from 14 to 70. The WEMWBS has been used in caregivers of persons with dementia (Orgeta, Lo Sterzo, & Orrell, 2013).
Change in the quality of life (WHO-Quality of Life BREF) score | Baseline (Visit 2/Week 1), Post-Intervention (Visit 3/Week 7)
  This 26-item questionnaire assesses quality of life across four domains: physical, psychological, social, and environmental ("Development of the World Health Organization WHOQOL-BREF Quality of Life Assessment," 1998) using a 5-point scale. It has been used in older adults, patients with dementia, and caregivers of Alzheimer's patients (Danucalov, Kozasa, Afonso, Galduroz, & Leite, 2017; von Steinbüchel, Lischetzke, Gurny, & Eid, 2006).
Change in the Sleep Disturbance score | Baseline (Visit 2/Week 1), Post-Intervention (Visit 3/Week 7)
  The PROMIS® (Patient-Reported Outcomes Measurement Information System) Sleep disturbance 8a is an 8-item self-rated index of sleep quality and sleep habits during the last seven days (Full, Malhotra, Crist, Moran, & Kerr, 2019). Higher values correspond to greater levels of sleep disturbance.
Change in the Multifactorial Memory Questionnaire (MMQ)-Ability scale score | Baseline (Visit 2/Week 1), Post-Intervention (Visit 3/Week 7)
  MMQ-Ability scale is a subscale of the MMQ that provides a measure of self-perception of everyday memory ability over the past two weeks, using 18 items rated on a 5-point scale ranging from "strongly agree" to "strongly disagree". High total scores indicate higher perceived ability. The MMQ was designed to be used in clinical assessment and interventions (Troyer & Rich, 2002), has been normed on older adults, and used with individuals with mild cognitive impairment (Kinsella et al., 2009; Troyer & Rich, 2002).
Change in the Multifactorial Memory Questionnaire (MMQ)-Satisfaction scale score | Baseline (Visit 2/Week 1), Post-Intervention (Visit 3/Week 7)
  The MMQ-Satisfaction scale evaluates overall concern or satisfaction with one's memory over the past two weeks using 18 items rated on a 5-point scale, ranging from "strongly agree" to "strongly disagree". High total scores indicate higher satisfaction. The MMQ was designed to be used in clinical assessment and interventions (Troyer & Rich, 2002), has been normed on older adults, and used with individuals with mild cognitive impairment (Kinsella et al., 2009; Troyer & Rich, 2002).
Change in the Conor-Davidson Resilience Scale (CD-RISC) score | Baseline (Visit 2/Week 1), Post-Intervention (Visit 3/Week 7)
  The 10-item Conor-Davidson Resilience Scale is a self-administered questionnaire that evaluates an individual's resilience over the past month. Respondents rate their agreement on 10 items on a scale from 0 (not true at all) to 4 (true nearly all the time). The final score is calculated by summing all the items (Campbell-Sills & Stein, 2007), with higher scores reflecting greater resilience.
10-item Burden Scale for Family Caregivers (BSFC-s) | Baseline (Visit 2/Week 1), Post-Intervention (Visit 3/Week 7)
  The BSFC-s is a self-administered 10-item scale designed to measure the subjective burden felt by informal caregivers (Graessel, Berth, Lichte, & Grau, 2014). Respondents rate their agreement on 10 items on a 4 point scale, from "strongly disagree" to "strongly agree". Higher total scores indicate greater subjective burden. This measure will be administered to the caregivers group only.
Average hours of technical support per person | Intervention period (6 weeks)
  Calls for technical assistance to study staff will be logged to estimate the amount of technical assistance required during a six week intervention. The average total hours per person spent will be calculated for each group and condition.
Change in visual working memory | Baseline (Visit 2/Week 1), Post-Intervention (Visit 3/Week 7)
  A modified Sternberg-type visual memory task will be used to evaluate effects on memory. Participants will view two faces shown one after another and will be asked to remember the faces and the order in which they were shown. After a brief retention interval (2 s), a number '1' or '2' will cue participants to recall the first or second face. A probe face will then appear and participants will indicate with a "Yes" or "No" whether the probe face matched the cued face. Both reaction time and accuracy will be used to evaluate memory performance.
Change in visual attention | Baseline (Visit 2/Week 1), Post-Intervention (Visit 3/Week 7)
  Attention will be measured using a variation of the attentional field of view task (Sekuler, Bennett, & Mamelak, 2000). In the focused-central condition, participants need to report which one of four letters was briefly flashed in the centre of the screen. In the focused-peripheral condition, participants report in which quadrant a small white circle was flashed in the periphery. In the divided-attention condition, participants report which letter was presented in the centre of the screen and which quadrant contained a flash in the periphery. The duration of the visual stimuli is varied to determine the minimum duration required to achieve a threshold level of performance. The ratio of duration thresholds in the focused and divided conditions for both tasks is the measure of performance of interest.
Change in event-related potentials in the auditory oddball task | Baseline (Visit 2/Week 1), Post-Intervention (Visit 3/Week 7)
  Three types of tones (frequent 1000 Hz tone, rare 1700 Hz target tone, and a rare 400 Hz deviant tone) will be played at random intermittent intervals. Participants will be asked to press a button as soon as the target tone is heard and not do anything for the other tones. EEG data will be recorded with the MUSE headband. The amplitude and latency of the N2 and P3 components of the event-related potentials time-locked to the three stimuli types will be analyzed.
Toronto Mindfulness Scale (TMS) | Intervention period (6 weeks)
  The TMS is a 13-item instrument assessing participants' mindfulness state immediately following an activity (Lau et al., 2006). Respondents rate their agreement with 13 statements on a 5-point scale, from "not at all" to "very much"; higher total scores correspond to greater levels of state mindfulness. Participants will complete this questionnaire once a week immediately following one of their meditation sessions. This scale will be used to examine how the quality of mindfulness changes across the six weeks of the intervention.
Change in the Credibility/Expectancy Questionnaire Score | Baseline (Visit 2/Week 1), Post-Intervention (Visit 3/Week 7)
  This questionnaire measures treatment expectancy and rationale credibility (Devilly & Borkovec, 2000). It has been used in dementia caregivers and older adults in the context of mindfulness meditation interventions (Oken et al., 2010; Wahbeh, Goodrich, & Oken, 2016). This scale will be used to assess whether participants in the two intervention arms have similar expectations and to examine whether expectations or credibility change from pre- to post- intervention.
Retention rate | Post-intervention visit (Visit 3/Week 7)
  The retention rate will be quantified as the proportion of participants enrolled in the study who complete the post-intervention assessment visit (Visit 3). This is a feasibility outcome variable.
Mean duration of meditation sessions | Intervention period (6 weeks)
  The average duration (in minutes) of completed meditation sessions will be obtained for each participant to evaluate adherence to the intervention schedule. This is an acceptability outcome variable.
Study acceptability score | Post-intervention visit (Visit 3, Week 7)
  Study acceptability will be evaluated with a single-item question 'how satisfied are you with the meditation intervention study you just took part in', with a rating from 1 (unsatisfied) to 9 (very satisfied). Additional items in a custom-made end-of-study user feedback survey will be used to provide more insight on the acceptability of the meditation technology and the study itself.
Change in EEG features during meditation | Intervention period (6 weeks)
  Participants' raw EEG data will be recorded with the MUSE headband throughout all meditation sessions. The EEG power spectrum within each session be quantified with the average power at classically defined frequency bands, alpha power asymmetry, peak alpha frequency, and the slope of the aperiodic signal.
Change in resting state EEG features with eyes open | Baseline (Visit 2/Week 1), Post-Intervention (Visit 3/Week 7)
  EEG data will be recorded with the Muse headband while participants are asked to sit still while looking at a fixation point on the screen for 2.5 minutes. This recording will be performed at the beginning and at the end of the assessment session. The EEG power spectral density will be quantified with the average power at classically defined frequency bands, alpha power asymmetry, peak alpha frequency, and the slope of the aperiodic signal.
Change in resting state EEG features with eyes closed | Baseline (Visit 2/Week 1), Post-Intervention (Visit 3/Week 7)
  EEG data will be recorded with the Muse headband while participants are asked to sit with their eyes closed for 2.5 minutes. This recording will be performed at the beginning and at the end of the assessment session. The EEG power spectral density will be quantified with the average power at classically defined frequency bands, alpha power asymmetry, peak alpha frequency, and the slope of the aperiodic signal.

OTHER OUTCOMES:
Change in far visual acuity | Baseline (Visit 2/Week 1), Post-Intervention (Visit 3/Week 7)
  Far visual acuity will be measured with the computerized FrACT test (Bach, 1996), which has been validated against standard acuity charts (Wesemann, 2002). The test presents letters one by one in the middle of the screen and asks participants to name them out loud, while the experimenter enters the letters on the keyboard. Each letter is presented at high contrast and an adaptive procedure changes the letter size in order to estimate the smallest readable letter.
Change in visual contrast sensitivity | Baseline (Visit 2/Week 1), Post-Intervention (Visit 3/Week 7)
  The computerized FrACT contrast sensitivity test (Bach, 1996) presents participants with a Landolt C in one of four orientations (up, down, left, or right) and participants are asked to indicate the direction where the C is pointing.

CONTACTS AND LOCATIONS:
Overall Officials: Allison B Sekuler, PhD, Principal Investigator — Baycrest; Morris Freedman, MD, FRCPC, Principal Investigator — Baycrest
Locations (1):
- Baycrest, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD that will be included in publications will be made available to other researchers. The dissemination platform is yet to be decided.
Supporting Information: Study Protocol
Time Frame: The data will become available at the time of publication of the articles and will remain accessible indefinitely.

REFERENCES:
- [Background] Anthony-Bergstone CR, Zarit SH, Gatz M. Symptoms of psychological distress among caregivers of dementia patients. Psychol Aging. 1988 Sep;3(3):245-8. doi: 10.1037//0882-7974.3.3.245. PMID 3268265
- [Background] Atchley R, Klee D, Memmott T, Goodrich E, Wahbeh H, Oken B. Event-related potential correlates of mindfulness meditation competence. Neuroscience. 2016 Apr 21;320:83-92. doi: 10.1016/j.neuroscience.2016.01.051. Epub 2016 Feb 3. PMID 26850995
- [Background] Bach M. The Freiburg Visual Acuity test--automatic measurement of visual acuity. Optom Vis Sci. 1996 Jan;73(1):49-53. doi: 10.1097/00006324-199601000-00008. PMID 8867682
- [Background] Campbell-Sills L, Stein MB. Psychometric analysis and refinement of the Connor-davidson Resilience Scale (CD-RISC): Validation of a 10-item measure of resilience. J Trauma Stress. 2007 Dec;20(6):1019-28. doi: 10.1002/jts.20271. PMID 18157881
- [Background] Chan JS, Kaiser J, Brandl M, Matura S, Prvulovic D, Hogan MJ, Naumer MJ. Expanded temporal binding windows in people with mild cognitive impairment. Curr Alzheimer Res. 2015;12(1):61-8. doi: 10.2174/1567205012666141218124744. PMID 25523426
- [Background] Danucalov MA, Kozasa EH, Afonso RF, Galduroz JC, Leite JR. Yoga and compassion meditation program improve quality of life and self-compassion in family caregivers of Alzheimer's disease patients: A randomized controlled trial. Geriatr Gerontol Int. 2017 Jan;17(1):85-91. doi: 10.1111/ggi.12675. Epub 2015 Dec 21. PMID 26685923
- [Background] Deeken F, Hausler A, Nordheim J, Rapp M, Knoll N, Rieckmann N. Psychometric properties of the Perceived Stress Scale in a sample of German dementia patients and their caregivers. Int Psychogeriatr. 2018 Jan;30(1):39-47. doi: 10.1017/S1041610217001387. Epub 2017 Jul 24. PMID 28737120
- [Background] Derogatis, L. R. (2001). BSI 18, Brief Symptom Inventory 18: Administration, scoring and procedures manual. NCS Pearson, Incorporated.
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Ezzati A, Jiang J, Katz MJ, Sliwinski MJ, Zimmerman ME, Lipton RB. Validation of the Perceived Stress Scale in a community sample of older adults. Int J Geriatr Psychiatry. 2014 Jun;29(6):645-52. doi: 10.1002/gps.4049. Epub 2013 Dec 3. PMID 24302253
- [Background] Full KM, Malhotra A, Crist K, Moran K, Kerr J. Assessing psychometric properties of the PROMIS Sleep Disturbance Scale in older adults in independent-living and continuing care retirement communities. Sleep Health. 2019 Feb;5(1):18-22. doi: 10.1016/j.sleh.2018.09.003. Epub 2018 Oct 28. PMID 30670160
- [Background] Graessel E, Berth H, Lichte T, Grau H. Subjective caregiver burden: validity of the 10-item short version of the Burden Scale for Family Caregivers BSFC-s. BMC Geriatr. 2014 Feb 20;14:23. doi: 10.1186/1471-2318-14-23. PMID 24555474
- [Background] Kinsella GJ, Mullaly E, Rand E, Ong B, Burton C, Price S, Phillips M, Storey E. Early intervention for mild cognitive impairment: a randomised controlled trial. J Neurol Neurosurg Psychiatry. 2009 Jul;80(7):730-6. doi: 10.1136/jnnp.2008.148346. Epub 2009 Mar 29. PMID 19332424
- [Background] Lau MA, Bishop SR, Segal ZV, Buis T, Anderson ND, Carlson L, Shapiro S, Carmody J, Abbey S, Devins G. The Toronto Mindfulness Scale: development and validation. J Clin Psychol. 2006 Dec;62(12):1445-67. doi: 10.1002/jclp.20326. PMID 17019673
- [Background] Levinson DB, Stoll EL, Kindy SD, Merry HL, Davidson RJ. A mind you can count on: validating breath counting as a behavioral measure of mindfulness. Front Psychol. 2014 Oct 24;5:1202. doi: 10.3389/fpsyg.2014.01202. eCollection 2014. PMID 25386148
- [Background] Milz P, Faber PL, Lehmann D, Kochi K, Pascual-Marqui RD. sLORETA intracortical lagged coherence during breath counting in meditation-naive participants. Front Hum Neurosci. 2014 May 15;8:303. doi: 10.3389/fnhum.2014.00303. eCollection 2014. PMID 24860483
- [Background] Orgeta V, Lo Sterzo E, Orrell M. Assessing mental well-being in family carers of people with dementia using the Warwick-Edinburgh Mental Well-Being Scale. Int Psychogeriatr. 2013 Sep;25(9):1443-51. doi: 10.1017/S1041610213000835. Epub 2013 Jun 19. PMID 23777581
- [Background] Petkus AJ, Gum AM, Small B, Malcarne VL, Stein MB, Wetherell JL. Evaluation of the factor structure and psychometric properties of the Brief Symptom Inventory-18 with homebound older adults. Int J Geriatr Psychiatry. 2010 Jun;25(6):578-87. doi: 10.1002/gps.2377. PMID 20013879
- [Background] Segal DL, Coolidge FL, Cahill BS, O'Riley AA. Psychometric properties of the Beck Depression Inventory II (BDI-II) among community-dwelling older adults. Behav Modif. 2008 Jan;32(1):3-20. doi: 10.1177/0145445507303833. PMID 18096969
- [Background] Sekuler AB, Bennett PJ, Mamelak M. Effects of aging on the useful field of view. Exp Aging Res. 2000 Apr-Jun;26(2):103-20. doi: 10.1080/036107300243588. PMID 10755218
- [Background] Steer RA, Brown GK, Beck AT, Sanderson WC. Mean Beck Depression Inventory-II scores by severity of major depressive episode. Psychol Rep. 2001 Jun;88(3 Pt 2):1075-6. doi: 10.2466/pr0.2001.88.3c.1075. PMID 11597055
- [Background] Takai M, Takahashi M, Iwamitsu Y, Ando N, Okazaki S, Nakajima K, Oishi S, Miyaoka H. The experience of burnout among home caregivers of patients with dementia: relations to depression and quality of life. Arch Gerontol Geriatr. 2009 Jul-Aug;49(1):e1-5. doi: 10.1016/j.archger.2008.07.002. Epub 2008 Aug 13. PMID 18703239
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Background] Troyer AK, Rich JB. Psychometric properties of a new metamemory questionnaire for older adults. J Gerontol B Psychol Sci Soc Sci. 2002 Jan;57(1):P19-27. doi: 10.1093/geronb/57.1.p19. PMID 11773220
- [Background] von Steinbuchel N, Lischetzke T, Gurny M, Eid M. Assessing quality of life in older people: psychometric properties of the WHOQOL-BREF. Eur J Ageing. 2006 May 31;3(2):116-122. doi: 10.1007/s10433-006-0024-2. eCollection 2006 Jun. PMID 28794757
- [Background] Wesemann W. [Visual acuity measured via the Freiburg visual acuity test (FVT), Bailey Lovie chart and Landolt Ring chart]. Klin Monbl Augenheilkd. 2002 Sep;219(9):660-7. doi: 10.1055/s-2002-35168. German. PMID 12410466
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119